CLINICAL TRIAL: NCT02768168
Title: The Effects of Dezocine Pretreatment on Dexamethasone Induced Perineal Irritation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mz2016
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Effect
Keywords: Dezocine; Dexamethasone 21-phosphate; Pain; Pruritus
MeSH Terms: conditions — Pain; Pruritus | interventions — dezocine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group D (Experimental): 40 patients receive dezocine 0.1 mg/Kg
  Interventions: Drug: dezocine
- Group C (Placebo Comparator): 40 patients receive matching placebo （normal saline）
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: dezocine — receive dezocine 0.1 mg/kg
  Arms: Group D
Other: normal saline — receive matching placebo (equal volume of normal saline)
  Arms: Group C

SUMMARY:
The purpose of this study is to investigate the efficacy of dezocine pretreatment on dexamethasone 21-phosphate induced perineal irritation (include pian and pruritus).

DETAILED DESCRIPTION:
Dexamethasone is a synthetic glucocorticoid, which may cause perineal irritation when given intravenously. The major clinical manifestations are pruritus and pain，and the incidence vary between 38%-71%. Some patients undergo spontaneous remission, while others develop into severe pain or pruritus. Dezocine, a new synthetic opiate agonist-antagonist, has been used for the treatment of pain and pruritus, but its role in relieving dexamethasone induced perineal irritation has not been studied yet. The aim of this study was to investigate the efficacy of dezocine pretreatment on dexamethasone induced perineal irritation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* ASA physical status I-II
* BMI 18-24.5 kg/m2

Exclusion Criteria:

* On regular use of analgesic
* Contraindication or allergy to steroid or dezocine
* Drug or alcohol abuse
* Diagnosed with paresthesia or mental diseases
* Communication disorders
* Pregnancy or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The occurrence of perineal irritation after the injection of dexamethasone 21-phosphate among Group D (40 patients receive dezocine 0.1 mg/Kg) and Group C (40 patients receive matching placebo) | In the first 3 min period after the injection of dexamethasone 21-phosphate phosphate

SECONDARY OUTCOMES:
The severity of perineal irritation after the injection of dexamethasone 21-phosphate among Group D (40 patients receive dezocine 0.1 mg/Kg) and Group C (40 patients receive matching placebo) | In the first 3 min period after the injection of dexamethasone 21-phosphate phosphate

OTHER OUTCOMES:
The duration of perineal irritation after the injection of dexamethasone 21-phosphate among Group D (40 patients receive dezocine 0.1 mg/Kg) and Group C (40 patients receive matching placebo) | In the first 3 min period after the injection of dexamethasone 21-phosphate phosphate

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Zheng, Principal Investigator — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No